CLINICAL TRIAL: NCT06139627
Title: Geriatric Assessment and Management (GAM) for Older Adults With Non-Small Cell Lung Cancer Receiving Chemotherapy Radiation Therapy (GAM-CRT)
Brief Title: Evaluation of Geriatric Assessment and Management for Older Adults With Non-small Cell Lung Cancer Receiving Chemotherapy Radiation Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23398; NCI-2023-07140 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23398 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2023-10-05; First posted 2023-11-18 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Lung Non-Small Cell Carcinoma; Stage III Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care; Specimen Handling; Geriatric Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (GA intervention) (Experimental): Patients complete a geriatric assessment. Patients and physicians receive the geriatric assessment summary and assessment-based recommendations, which are provided prior to beginning chemotherapy and radiation, at the midpoint of chemotherapy and radiation treatment, and at the end of treatment. Patients also undergo blood and stool sample collection during screening and on study.
  Interventions: Procedure: Biospecimen Collection; Other: Communication Intervention; Other: Comprehensive Geriatric Assessment; Other: Electronic Health Record Review; Other: Survey Administration
- Arm II (usual care) (Active Comparator): Patients complete a geriatric assessment, but information other than clinically significant cognitive impairment and depression is not provided to the oncology teams, per usual care. Patients also undergo blood and stool sample collection during screening and on study.
  Interventions: Other: Best Practice; Procedure: Biospecimen Collection; Other: Comprehensive Geriatric Assessment; Other: Electronic Health Record Review; Other: Survey Administration

INTERVENTIONS:
Other: Best Practice — Receive usual care
  Other Names: standard of care; standard therapy
  Arms: Arm II (usual care)
Procedure: Biospecimen Collection — Undergo blood and stool sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Communication Intervention — Receive GA assessment summary and assessment-based recommendations
  Arms: Arm I (GA intervention)
Other: Comprehensive Geriatric Assessment — Complete GA
Other: Electronic Health Record Review — Ancillary studies
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial tests how well a geriatric assessment (GA) with GA-directed treatment recommendations, compared to GA with usual care, works in identifying risk factors, reducing chemotherapy radiation toxicity and functional decline, and improving the overall quality of life in older patients with non-small cell lung cancer (NSCLC). Older patients with lung cancer undergoing chemotherapy are at an increased risk of adverse outcomes including treatment toxicity and functional and physical consequences. This makes it very challenging for the physicians to balance the benefits against the risk of chemotherapy in older cancer patients. A geriatric assessment may be useful in identifying risk factors for chemotherapy radiation toxicity. Communicating these geriatric assessment findings and assessment-based recommendations to a patient's treating physicians may help them make more informed decisions about treatment options for patients. Making treatment decisions using GA-based recommendations may reduce adverse events and improve outcomes in patients receiving treatment for NSCLC.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To demonstrate if providing a GA summary and recommendations for GA-directed interventions to oncology care teams decreases the proportion of older adults with unresectable, stage III NSCLC who experience any grade 3-5 non-hematologic toxicity from chemotherapy and radiation.

SECONDARY OBJECTIVES:

I. To demonstrate the differences between the intervention versus usual care group among:

Ia. Overall grade 3-5 toxicities; Ib. Patient-reported symptomatic toxicities as measured by Patient Reported Outcomes - Common Terminology Criteria for Adverse Events (PROCTCAE), Patient Reported Outcomes Measurement Information System - 10 (PROMIS-10); Ic. Implementation of GA recommendations; Id. GA outcomes including function (Activities of Daily Living/Instrumental Activities of Daily Living,), physical performance (Short Physical Performance Battery, 2 minute [min] walk, falls), polypharmacy (reduction in medication burden), mood (Geriatric Depression Scale 5/15 and PROMIS Anxiety short form 4a); Ie. Quality of life (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 [EORTC-QLQ-30]); If. Treatment sequencing (concurrent versus sequential) and completion, hospitalizations/emergency department (ED) rates.

EXPLORATORY OBJECTIVE:

I. To explore microbial diversity and blood components at baseline, and at 6 months from treatment initiation as a potential biomarker of treatment-related toxicity and disease response.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients complete a geriatric assessment. Patients and physicians receive the geriatric assessment summary and assessment-based recommendations, which are provided prior to beginning chemotherapy and radiation, at the midpoint of chemotherapy and radiation treatment, and at the end of treatment. Patients also undergo blood and stool sample collection during screening and on study.

ARM II: Patients complete a geriatric assessment, but information other than clinically significant cognitive impairment and depression is not provided to the oncology teams, per usual care. Patients also undergo blood and stool sample collection during screening and on study.

After completion of study intervention, patients are followed up at 4-6 weeks, 10-14 weeks, and 20-26 weeks after baseline.

ELIGIBILITY:
Inclusion Criteria:

* ONCOLOGY PHYSICIANS INCLUSION:
* Oncology physicians must work at the participating site with no plans to leave that site or retire at the time of enrollment into the study
* PATIENTS INCLUSION:
* Any patient with unresectable non-small cell lung cancer diagnosis who is 60 years of age or older and must be treated at the participating site
* Clinical staging without pathological confirmation of nodal disease is allowed
* Plan to start a new cancer treatment regimen within 4-6 weeks from time of baseline study visit. The treatment regimen is up to the discretion of the treating oncology physician. The regimen must include a chemotherapy drug or other agents that have similar prevalence of toxicity. This can be either concurrent or sequential with radiation therapy
* Chemotherapy will be defined as cytotoxic drugs; in addition, agents (e.g., monoclonal antibodies and targeted agents) will be allowed. Given the rapidly changing landscape of new drugs for cancer, the study team led by the principal investigator (PI) will update the list accordingly after reviewing the toxicity profile of new therapies
* Patients who are receiving approved cancer treatment in combination or sequentially with radiation including hypo fractionated radiation (45-60Gy in 15-20 fractions) are eligible
* Those patients with oligometastatic disease having only one site and one lesion outside of the radiation field will be eligible. Examples include a solitary brain metastasis (met), contralateral lung nodule or an adrenal metastatic site
* A patient may also be enrolled on a treatment trial and participate in this study, if all other inclusion and exclusion criteria are met
* Able to provide informed consent, or if the oncology physician determines the patient to not have decision-making capacity, a patient-designated health care proxy (or authorized representative per institutional policies) must sign consent by the baseline visit
* Participant or healthcare proxy has adequate understanding of the English language (preferred) because not all GA measures have been validated in other languages. Study team should be contacted for any participants with other preferred languages including Spanish and Mandarin. Inclusion of these participants will depend upon the availability of the translators and their ability to accurately translate the measures as approved by the local Institutional Review Board (IRB)

Exclusion Criteria:

* PATIENTS EXCLUSION:
* Have surgery planned within 3 months of approach date. Patients who have previously received surgery are eligible
* Presence of symptomatic brain metastases (if more than one) at time of study consent process. Patients with history of treated brain metastases or small indeterminate lesions (< 1cm) are eligible if they are not symptomatic at the time of study enrollment
* More than one metastatic site: Examples: brain and adrenal, adrenal and liver

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2026-07-19 (Estimated); Study Completion 2026-07-19 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade 3-5 non-hematologic toxicities | At 6 months from treatment initiation
  Will be assessed by National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (NCI CTCAE v 5.0) for grade 3-5 non-hematologic toxicities. Chi-square test will be used to compare proportion of patients with grade 3-5 non-hematologic toxicity between two arms at 6 months after treatment initiation.

SECONDARY OUTCOMES:
Overall grade 3 to 5 toxicities | At 6 months from treatment initiation
  Will be assessed by National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (NCI CTCAE v 5.0) for grade 3-5 toxicities. Chi-square test will be used to compare proportion of patients with grade 3-5 toxicities between two arms at 6 months after treatment initiation.
Patient-reported symptomatic toxicities | At 6 months from treatment initiation
  Will be assessed by the Patient Reported Outcome version of the Common Terminology Criteria for Adverse Events and Patient Reported Outcomes Measurement Information System (PROMIS)-10. Chi-square test or fisher's exact test will be used to examine the difference between the two arms.
Function | At 6 months from treatment initiation
  Will be assessed by activities of daily living/instrumental activities of daily living. T test Chi-square test or fisher's exact test will be used to examine the difference between the two arms.
Physical performance -SPPB | At 6 months from treatment initiation
  Will be assessed by the short physical performance battery (SPPB) which is scored according to instruction, range from 0 to 12), T test, Chi-square test or fisher's exact test will be used to examine the difference between the two arms.
Physical performance - 2 minute walking | At 6 months from treatment initiation
  Will be assessed by 2 minute walking test (meters). T test, Chi-square test or fisher's exact test will be used to examine the difference between the two arms.
Physical performance - number of falls | At 6 months from treatment initiation
  Will be assessed by number of falls (count number). T test, Chi-square test or fisher's exact test will be used to examine the difference between the two arms.
Polypharmacy | At 3 months from treatment initiation
  Will be assessed by the reduction in medication burden. Chi-square test or fisher's exact test will be used to examine the difference between the two arms.
Mood - GDS | At 6 months from treatment initiation
  Will be assessed by the Geriatric Depression Scale (GDS) 5/15 (scored according to guideline).
  T test, Chi-square test or fisher's exact test will be used to examine the difference between the two arms.
Mood - Anxiety | At 6 months from treatment initiation
  Will be assessed by PROMIS anxiety (scored according to guideline). T test, Chi-square test or fisher's exact test will be used to examine the difference between the two arms.
Quality of life | At 6 months from treatment initiation
  Will be assessed by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 scored according to guideline.
  T test, Chi-square test or fisher's exact test will be used to examine the difference between the two arms.
Treatment completion rates | At 6 months from treatment initiation
  Chi-square test or fisher's exact test will be used to examine the difference between the two arms.
Hospitalizations/emergency department visit rates | At 6 months from treatment initiation
  Chi-square test or fisher's exact test will be used to examine the difference between the two arms.
Incidence of adverse events from durvalumab | After completion of adjuvant treatment (12 months)
  Chi-square test or fisher's exact test will be used to examine the difference between the two arms.

CONTACTS AND LOCATIONS:
Overall Officials: Arya Amini, Principal Investigator — City of Hope Medical Center
Locations (3):
- United States (3):
  - City of Hope Medical Center, Duarte, California
  - University of Rochester, Rochester, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio